CLINICAL TRIAL: NCT03110965
Title: Yoga in the Treatment of Adolescent Idiopathic and Degenerative Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manhattan Physical Medicine and Rehabilitation, LLP (Other)
Responsible Party: Principal Investigator, Loren M. Fishman,MD, Assistant Clinical Professor, Columbia University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MANHATTANPMR
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Scoliosis; Scoliosis Idiopathic
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Patient's change in previous X-ray compared with baseline, and baseline compared with X-ray done 4-10 months later
Masking Description: Radiologists are unaware of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients will have an X-ray before beginning to do one or two yoga poses daily for 4 - 10 months. After that period, they will have a second X-ray.
  Interventions: Behavioral: Yoga poses

INTERVENTIONS:
Behavioral: Yoga poses — Patients are asked to perform one or two yoga poses daily for 4-10 months

SUMMARY:
The effect of two isometric exercises is measured on Cobb angles from films taken 4-10 months apart.

DETAILED DESCRIPTION:
The investigators obtained baseline Cobb angles on simple and complex curves, and collected previous, earlier studies of each adolescent idiopathic and degenerative scoliosis patient. The investigators then taught them to do the side-plank pose with the convex side of lumbar and thoracolumbar scoliotic curves downward, and a slightly altered version of the the half moon pose of yoga with the convex side of thoracic and cervicothoracic curves downward. The half moon pose was altered in that a belt was looped around the horizontal leg's foot, and held in a vertically extended upper arm's hand, and pulled tightly in that vertical position.

Each pose was held as long as the patient could at least once daily.

Cobb angles were again measured in films taken 4-10 months later.

ELIGIBILITY:
Inclusion Criteria:

* Scoliosis
* Willingness to do pose at least once daily for 4 -10 months
* Willingness to have a second X-ray 4-10 months after starting to do pose

Exclusion Criteria:

* Neuromuscular disease
* Previous Spinal surgery
* Pregnancy

Ages: 6 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Cobb angle | 4 - 10 months
  Baseline scoliotic curve - scoliotic curve measured after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Loren M Fishman, MD, Principal Investigator — Columbia Medical School
Locations (1):
- Manhattan Physical Medicine and Rehabilitation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No